CLINICAL TRIAL: NCT05312853
Title: Evaluating the Diagnostic and Predictive Value of Non-invasive Tests (NITs) on the Progression of Chronic Liver Disease.
Acronym: NITOutcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Boehringer Ingelheim (Industry); Nordic Bioscience A/S (Industry)
Responsible Party: Principal Investigator, Jörn M. Schattenberg, Prof. Dr., Johannes Gutenberg University Mainz
Other Study IDs: 21-02552
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. 3 x 5mls into EDTA (purple) Vacutainer blood tubes - used for plasma collection for subsequent biomarker or metabolomic/proteomic/miRNA/cell-free DNA analyses and cellular DNA extraction.
  2. 4 x 5mls (or 2 x 10mls) into GOLD top SST Vacutainer tubes (serum) - used for serum collection for subsequent biomarker or metabolomic/proteomic/miRNA/cell-free DNA analyses. [Note: RED top Vacutainer tubes (serum) may be substituted if GOLD tubes are not available locally].
  3. 1 x 5mls into PAX tube for RNA preservation - for peripheral blood RNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objective is to study the relevance of non-invasive test (NITs) in predicting disease stage (diagnostic biomarker) and outcome (predictive biomarker) in patients with suspected or established liver disease and cirrhosis.

DETAILED DESCRIPTION:
Non-invasive tests (NITs) may complement and even reduce the need for liver biopsy in the diagnosis and follow up care of patients with chronic liver disease (CLD). NITs either include serum biomarkers (direct or indirect) or ultrasound-based tests, including vibration controlled transient elastography (VCTE), or a combination of both incorporated into several surrogate scores.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Clinically suspected chronic liver disease based on any of:

   1. Patient with historical liver biopsy providing histological evidence of any liver disease or,
   2. Patient undergoing liver biopsy for suspected chronic liver disease with biochemical and/or radiological findings consistent with liver disease or,
   3. Patient with clinical and radiological evidence of cirrhosis (in absence of an alternative aetiology)
   4. Patients with metabolic risk factors predisposing to CLD

Exclusion Criteria:

1. Refusal or inability (lack of capacity) to give informed consent.
2. Age < 18 years
3. Pregnancy
4. An active malignancy.
5. Life expectation of < 5 years.
6. Patients not meeting inclusion criteria or judged by the investigator to be unsuitable for inclusion in the study.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be patients (aged ≥18 years) with risk factors for chronic liver disease recruited at the I. Department of Medicine of the University Medical Center Mainz in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2034-04-15 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years
  The primary objective of this observational study is to assemble a cohort of well-characterised patients with chronic liver disease (CLD) and to collect associated clinical information, biological samples and imaging data for cross-sectional and longitudinal analyses in order to robustly validate diagnostic and predictive non-invasive tests (NITs) for the diagnosis, risk assessment (prognosis) and monitoring of patients with liver disease.
  The primary outcome will be overall survival.

SECONDARY OUTCOMES:
Liver-related events | 10 years
  Longitudinal correlation of phenotype with liver -related outcome and transplant-free survival.

OTHER OUTCOMES:
Impact of liver disease on Quality of Life and Symptom-burden | 5 years
  * Study of symptom burden in patients with CLD (Quality of Life).
  * Study the underlying pathogenic processes contributing to disease progression in CLD

CONTACTS AND LOCATIONS:
Overall Officials: Joern Schattenberg, Prof. Dr., Principal Investigator — Hepatology
Locations (1):
- University Medical Center of the Johannes Gutenber Univeristy, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No
The data and samples held by the Registry will be the property of the PI Prof. Jörn Schattenberg and the University Medical Center Mainz. Publication will be the responsibility of the PI in line with the polices established with partners in separate agreements and the requirements of the European Commission for open access publication. Scientific contributions will be duly and appropriately acknowledged in line with the 'Uniform Requirements for Articles Submitted to Biomedical Journals' produced by the Committee of Medical Journal Editors (2008).